CLINICAL TRIAL: NCT05981768
Title: A Phase 1 Study to Investigate the Effect of Food on the Bioavailability of a Single Cytisinicline 3 mg Tablet and Evaluation of the Pharmacokinetics of Multiple 3 mg Doses (Three Times Daily) in Healthy Adult Smokers
Brief Title: Study to Evaluate Effect of Food on Bioavailability of Single 3 mg Tablet and Pharmacokinetics (PK) of Multiple 3 mg Doses in Healthy Adult Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ACH-CYT-11
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Cytisinicline 3 mg Once Daily (QD), Fasting (Experimental): 3 mg cytisinicline tablet administered in the morning, between 7:00 and 9:00 AM, in fasting conditions on Day 1 (Period 1) or Day 3 (Period 2). Participants will fast overnight for at least 10 hours before cytisinicline administration and will continue to fast for 4 hours after dosing.
  Interventions: Drug: Cytisinicline
- Part 1: Cytisinicline 3 mg QD, Fed (Experimental): 3 mg cytisinicline tablet administered in the morning, between 7:00 and 9:00 AM, in fed conditions on Day 1 (Period 1) or Day 3 (Period 2). After an overnight fasting of at least 10 hours, participants will consume a standard high-fat-high-calorie meal within 30 minutes. Cytisinicline will be administered with 240 mL of water within 5 minutes after completion of the meal.
  Interventions: Drug: Cytisinicline
- Part 2: Cytisinicline 3 mg 3 Times Daily (TID) (Experimental): 3 mg cytisinicline tablet administered TID each day on Day 5 to 8 (Period 3) as follows: Dose 1 will be administered in the morning between 7:00 and 9:00 AM,; Dose 2 at 5 hours (±10 minutes) after Dose 1; Dose 3 at 5 hours (±10 minutes) after Dose 2. Cytisinicline will be administered on an empty stomach (cytisinicline given at least 2 hours before food or 1 hour after food).
  Interventions: Drug: Cytisinicline

INTERVENTIONS:
Drug: Cytisinicline — film-coated oral tablets containing 3 mg cytisinicline
  Other Names: Cytisine

SUMMARY:
To assess the effect of food on the bioavailability of 3 mg cytisinicline following single-dose administration, and to evaluate the PK profile of 3 mg cytisinicline TID following multiple days of administration during Days 5-8.

ELIGIBILITY:
Inclusion Criteria:

1. Free written informed consent prior to any procedure required by the study.
2. Willingness to accept and comply with all study procedures and restrictions.
3. Male or female subject ≥ 18 years, at the date of signing the informed consent.
4. Regular moderate combustible cigarette smokers (self-reported average of at least 10 cigarettes per day).
5. Body mass index (BMI) of 18.0 to 30.0 kg/m^2, inclusive.
6. Healthy subject, based on medical history, physical examination, vital signs, ECG and clinical laboratory tests.
7. Negative test results for anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV-1Ab and anti-HIV-2Ab), Hepatitis B surface antigen (HBsAg) and anti-hepatitis C virus antibodies (anti-HCVAb).
8. A female subject is eligible if she also meets one of the following criteria:

   1. is of non-childbearing potential (underwent a permanent sterilization method [eg, hysterectomy, bilateral salpingectomy or bilateral oophorectomy], is clinically diagnosed infertile, or is in a post-menopausal state); or
   2. is of childbearing potential and agrees to use an accepted contraceptive method from at least 4 weeks prior to admission and until at least 4 weeks after the last dose administration (Day 8).

Exclusion Criteria:

AT SCREENING

1. Known hypersensitivity/allergic reaction to cytisinicline or any of the excipients.
2. Known severe hypersensitivity reaction to any other drug.
3. Any medical condition (eg, gastrointestinal, renal or hepatic, including peptic ulcer, inflammatory bowel disease or pancreatitis) or surgical condition (eg, cholecystectomy, gastrectomy) that may affect drug pharmacokinetics (absorption, distribution, metabolism or excretion) or subject safety.
4. Stroke or acute myocardial infarction within the previous 3 months.
5. History of hyperthyroidism.
6. History of psychosis or of a psychotic event.
7. Estimated renal creatinine clearance (CLCr) below the lower limit of the normal range (ie, 90-120 mL/min/1.73 m^2 for males and 80-110 mL/min/1.73 m^2 for females), based on creatinine clearance calculation by the Cockcroft-Gault formula and normalized to an average body surface area of 1.73 m^2.
8. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) above the upper limit of the normal (ULN) range.
9. Positive result in urine drugs-of-abuse or ethanol tests at Screening.
10. Excessive caffeine consumption, defined as ≥ 800 mg per day.
11. Veins unsuitable for intravenous puncture on either arm (eg, veins that are difficult to locate, access or puncture; veins with a tendency to rupture during or after puncture).
12. Participation in any clinical trial within the previous 2 months.
13. Use of any smoking cessation medications such as cytisinicline, bupropion, varenicline, nortriptyline, or any nicotine replacement therapy (NRT; eg, nicotine patch, nicotine chewing gum, or electronic cigarettes) in the previous 8 weeks.
14. Participation in more than 2 clinical trials within the previous 12 months.
15. Blood donation or significant blood loss (≥ 450 mL) due to any reason or had plasmapheresis within the previous 2 months.
16. Female subjects who are lactating or pregnant by serum pregnancy test.
17. Any other condition that the investigator considers the subject to be unsuitable for the study.

    AT ADMISSION
18. Any recent disease or condition or treatment that, according to the investigator, would put the subject at undue risk due to study participation or occurred at a time frame in which may interfere with the pharmacokinetics of study drug.
19. Use of any medicinal products, prescription and non-prescription (including vitamins, food supplements, herbal supplements [including St John's Wort]), in the previous 2 weeks, unless in the investigator's opinion the medication does not interfere with the pharmacokinetics of study drug or compromise subject safety.

    NOTE: The use of topical products without systemic absorption, acetaminophen (paracetamol) at doses of ≤ 2 grams/day, and hormonal contraceptives are acceptable.
20. Use of any smoking cessation medications (eg, cytisinicline, bupropion, varenicline, nortriptyline, or any NRT eg, nicotine patch, nicotine chewing gum, or electronic cigarettes) since Screening.
21. Positive result in drugs-of-abuse or ethanol tests.
22. If female, positive pregnancy test in urine.
23. Any other condition that the investigator considers to render the subject unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Time of Maximum Observed Plasma Concentration (Tmax) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Time Point Prior to the First Quantifiable Concentration (Tlag) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Time of Last Quantifiable Observed Concentration (Tlast) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Area Under Plasma Concentration-Time Curve (AUC) Over the Dosing Interval (AUC0-τ) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
AUC From Time of Dosing (t=0h) to the Time of the Last Quantifiable Concentration (AUC0-t) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Total AUC Extrapolated to Infinity (AUC0-∞) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Percentage of AUC0-∞ Due to Extrapolation From the Time of the Last Quantifiable Concentration (Tlast) to Infinity (%AUCextrap) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Apparent Terminal Elimination Rate Constant (λz) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Apparent Terminal Elimination Half-Life (t1/2) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Apparent Clearance (CL/F) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Apparent Volume of Distribution (V/F) | Day 1 (Period 1) and Day 3 (Period 2): pre-dose and up to 24 hours post-dose
Pre-dose Plasma Concentration (Ctrough) for Dose 1, Dose 2 and Dose 3 | Days 5 to 8 (Period 3): pre-dose
Cmax for Dose 1, Dose 2 and Dose 3 | Days 5-7 (Period 3): predose, Day 8 (Period 3): pre-dose and up to 5 hours post-dose (Doses 1 and 2), predose and up to 24 hours post-dose (Dose 3)
Tmax for Dose 1, Dose 2 and Dose 3 | Days 5-7 (Period 3): predose, Day 8 (Period 3): pre-dose and up to 5 hours post-dose (Doses 1 and 2), predose and up to 24 hours post-dose (Dose 3)
AUC0-τ for Dose 1, Dose 2 and Dose 3 | Days 5-7 (Period 3): predose, Day 8 (Period 3): pre-dose and up to 5 hours post-dose (Doses 1 and 2), predose and up to 24 hours post-dose (Dose 3)
  τ=5 h for Dose 1 and Dose 2 and τ=24 h for Dose 3
Concentration Over the Dosing Interval (Cτ) for Dose 1, Dose 2 and Dose 3 | Days 5-7 (Period 3): predose, Day 8 (Period 3): pre-dose and up to 5 hours post-dose (Doses 1 and 2), predose and up to 24 hours post-dose (Dose 3)
  τ=5 h for Dose 1 and Dose 2 and τ=24 h for Dose 3
Apparent Terminal Elimination Half-Life Interval (t1/2) post Dose 3 | Day 8 (Period 3): up to 24 hours post-dose 3
Ratio of Cmax (R[Cmax]) | Day 1 (Period 1) or Day 3 (Period 2), Day 8 (Period 3): Dose 1 (up to 5 hours post-dose)
  Accumulation of cytisinicline following TID administration will be assessed by estimating R(Cmax), where R is the ratio of the pharmacokinetic parameter following administration of Dose 1 on Day 8 vs. single-dose administration under fasting conditions during Period 1 or 2.
Ratio of AUC0-τ (R[AUC0-τ]) | Day 1 (Period 1) or Day 3 (Period 2), Day 8 (Period 3): Dose 1 (up to 5 hours post-dose)
  Accumulation of cytisinicline following TID administration will be assessed by estimating R(AUC0-τ), where R is the ratio of the pharmacokinetic parameter following administration of Dose 1 on Day 8 vs. single-dose administration under fasting conditions during Period 1 or 2.
R(AUC0-τ/AUC0-∞) | Day 1 (Period 1) or Day 3 (Period 2), Day 8 (Period 3): Dose 1 (up to 5 hours post-dose)
  Time invariance will be assessed as R(AUC0-τ/AUC0-∞), where AUC0-τ is estimated on Day 8 Dose 1 and AUC0-∞ is estimated for the single-dose under fasting conditions during Period 1 or 2.
Time to Steady State | Days 5 to 8 (Period 3): pre-dose
  Time to steady state will be assessed by visual inspection of the Ctrough versus time plot.
Number of Participants With Treatment Emergent Adverse Events (AEs) | From first dose of study drug through the End-of Study Visit (Day 28-31)
Number of Participants With Clinically Significant Changes From Baseline in Electrocardiograms (ECG) | Baseline through Day 9
Number of Participants With Clinically Significant Changes From Baseline in Vital Signs | Baseline through Day 9
Number of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Tests | Baseline through Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fonseca, MD, Principal Investigator — Blue Clinical
Locations (1):
- BlueClinical Phase I, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No